CLINICAL TRIAL: NCT06211335
Title: Phase Ib Study of Losartan, Pembrolizumab and Stereotactic Body Radiation Therapy (SBRT) in Patients With Locoregionally Recurrent, Refractory, or Oligometastatic Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Losartan, Pembrolizumab and Stereotactic Body Radiation Therapy for the Treatment of Patients With Locally Recurrent, Refractory or Oligometastatic Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shyam S.D. Rao (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Shyam S.D. Rao, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC311; NCI-2023-10476 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC311 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Locally Recurrent Head and Neck Squamous Cell Carcinoma; Metastatic Head and Neck Squamous Cell Carcinoma; Refractory Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Losartan; pembrolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (losartan, SBRT, pembrolizumab) (Experimental): Patients receive losartan PO QD. One week later patients receive SBRT 2-3 times per week for approximately 2 weeks. Within 1 week of completing SBRT, patients receive pembrolizumab IV and repeat every 3 weeks. Treatment continues for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients undergo PET, tumor biopsy, and blood sample collection throughout the study.
  Interventions: Drug: Losartan; Biological: Pembrolizumab; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Losartan — Given PO
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; Keytruda; Lambrolizumab; MK-3475; Pembrolizumab Biosimilar BCD-201; SCH 900475
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase Ib trial tests the safety, side effects and how well losartan, pembrolizumab and stereotactic body radiation therapy (SBRT) for the treatment of patients with head and neck squamous cell carcinoma that has come back to nearby tissue or lymph node after a period of improvement (locally recurrent), that has not responded to previous treatment (refractory) or that has spread from where it first started to multiple other placed in the body (oligometastatic). Losartan is a drug used to treat high blood pressure that may enhance the effects of other cancer treatments such as immunotherapy and radiation. Immunotherapy with pembrolizumab may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. SBRT is a type of external radiation therapy that uses special equipment to position a patient and precisely deliver radiation to tumors in the body (except the brain). The total dose of radiation is divided into smaller doses given over several days. This type of radiation therapy helps spare normal tissue. Giving losartan, pembrolizumab and SBRT may work better in treating patients with locally recurrent, refractory or oligometastatic head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:I. Determine the safety and toxicity of losartan in combination with SBRT and subsequently pembrolizumab in patients with locally recurrent, refractory, or oligometastatic head and neck squamous cell carcinoma (HNSCC).

SECONDARY OBJECTIVES:I. Evaluate objective tumor response.II. Evaluate progression free survival (PFS). III. Evaluate duration of response.IV. Evaluate overall survival (OS).

OUTLINE:Patients receive losartan orally (PO) once daily (QD). One week later patients receive SBRT 2-3 times per week for approximately 2 weeks. Within 1 week of completing SBRT, patients receive pembrolizumab intravenously (IV) and repeat every 3 weeks. Treatment continues for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients undergo positron emission tomography (PET), tumor biopsy, and blood sample collection throughout the study.After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locoregionally recurrent, refractory, or oligometastatic (at most 4 lesions) squamous cell carcinoma of the head and neck not amenable to curative resection
* p16 status known for base of tongue, soft palate, and tonsil cancers
* Tumor amenable to sequential biopsies, and patients willing to undergo sequential tumor biopsies so long as the treating investigator considers them to be clinically safe
* Prior radiotherapy to the head and neck is allowed. Disease should be limited to up to 4 sites of active disease in the head and neck and/or distant metastatic sites if deemed safely treatable by physician, or adjacent sites treatable in single contiguous target volume with a recommended maximum total tumor dimension (GTV) of < 7.5 cm. However, larger volumes may be allowed after discussion with primary investigator (PI) and careful review of radiation dose constraints
* Prior systemic therapy is allowed. Patients with locoregional relapses where radiation alone would be indicated are allowed to enroll without prior systemic therapy
* Presence of measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) with a target on a computed tomography (CT) scan or magnetic resonance imaging (MRI) available for review
* Combined positive score (CPS) > 1%
* Age ≥ 18 years at time of consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
* Leukocytes ≥ 3 × 10^9/L
* Absolute neutrophil count ≥ 1.5 × 10^9/L
* Platelets ≥ 100 × 10^9/L
* Hemoglobin (Hgb) ≥ 9 g/dL, transfusions may be used to raise Hgb to ≥ 9 g/dL (no washout required)
* Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
* Aspartate transaminase (AST) / alanine transaminase (ALT) ≤ 2.5 × institutional ULN
* Creatinine within normal institutional limits OR creatinine clearance ≥ 30 mL/min/1.73 m^2 for patients with creatinine above institutional ULN
* The effects of losartan on the developing human fetus are unknown. For this reason, individuals of childbearing potential and male participants with partners of childbearing potential, must agree to use methods of contraception for the duration of study participation (including dosing interruptions) and for up to 3 months after last study treatment; or be surgically sterilized
* Ability to understand and willingness to sign and date the informed consent form
* Stated ability and willingness to adhere to the study visit schedule and protocol requirements

Exclusion Criteria:

* Nasopharyngeal carcinoma, salivary gland carcinoma or primary skin squamous cell carcinoma (SCC)
* Prior treatment with an anti-PD-1, anti-PD-L1, or anti-PD-L2 antibody
* Chemotherapy or other anti-cancer therapy within 3 weeks prior to study day 1
* Hypersensitivity to losartan or any component of the formulation
* Radiation therapy within 6 months prior to study day 1
* Patients with disease surrounding > 50% of the carotid
* Participant who has not recovered to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade ≤ 1 from an adverse event (AE) due to previous cancer therapeutics (i.e., chemotherapy, radiation therapy, biologic therapy, and/or experimental therapy) with the exception of alopecia
* Major surgery as assessed by the investigator (with the exception of diagnostic biopsy) within ≤ 28 days prior to study day 1 (patients must have completely recovered from any previous surgery prior to study day 1)
* Clinically significant bleeding ≤ 4 weeks prior to study day 1
* Requirement for parenteral antibiotics, or any active infection requiring parenteral antibiotic therapy within 4 weeks prior to study day 1
* Clinically significant or uncontrolled diabetes mellitus (hemoglobin A1C ≤ 8.5%). Patients with diabetes mellitus treated with aliskiren ≤ 7 days prior to study day 1 are excluded
* Active autoimmune disorders that have required systemic treatment with disease modifying agents, corticosteroids, or immunosuppressive drugs in the past 2 years are excluded. Patients with autoimmune disorder or well-managed or inactive autoimmune disorders, such as Hashimoto's thyroiditis, may be allowed at the discretion of the PI
* Current use of systemic corticosteroids equivalent to >10 mg of prednisone per day
* Current use of angiotensin receptor blockers (ARBs) or angiotensin converting enzyme (ACE) inhibitors for management of hypertension
* Clinically significant cardiovascular, pulmonary, endocrine, neurologic, gastrointestinal or genitourinary disease unrelated to underlying solid tumor that in the judgment of the investigator should preclude treatment with losartan
* Any other active malignancy except for low-risk prostate cancer previously treated or under active surveillance, uncomplicated and cured basal cell carcinoma, or squamous cell carcinoma of the skin within 5 years of study entry
* Known history of positive hepatitis C (HCV) antibody, hepatitis B (HBV) surface antigen (HbsAg and HBV core Ab positive), or human immunodeficiency virus (HIV) antibody results. Patients with positive antibody tests are eligible with negative viral loads
* Administration of live, attenuated vaccine ≤ 28 days prior to study day 1. Administration of inactivated flu vaccines is allowed
* Any prior treatment with losartan or other specific TGF-β-directed therapy
* Treatment with another investigational drug or device, or approved therapy for investigational use ≤ 28 days prior to study day 1, or if the half-life of the previous product is known, within 5 times the half-life prior to study day 1, whichever may be longer
* Pregnant or breast feeding
* Any condition that in the opinion of the investigator would interfere with the participant's safety, compliance while on trial, or understanding or rendering of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events | Up to 2 years
  Classified by severity and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 and summarized using descriptive statistics in participants treated with dosage of the agent selected in the safety run.

SECONDARY OUTCOMES:
Objective response rate | Up to 2 years
  Defined as stable disease, complete response (CR) or partial response (PR) on imaging assessed by Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Will be summarized using Kaplan-Meier curves and 95% confidence interval (CI). Median and range will be reported.
Progression free survival | From start of stereotactic body radiation therapy (SBRT) to local or distant progression or death due to any cause, up to 2 years
  According to RECIST 1.1. Will be summarized using Kaplan-Meier curves and 95% CI.
Duration of response | From CR or PR until progressive disease, death or last tumor assessment using RECIST 1.1, up to 2 years
  Median and range will be reported.
Overall survival | From the start of SBRT to death from any cause, up to 2 years
  Will be summarized using Kaplan-Meier curves and 95% CI.

CONTACTS AND LOCATIONS:
Overall Officials: Shyam S.D. Rao, MD, PhD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Colorado Denver | Anschutz Medical Campus, Aurora, Colorado